CLINICAL TRIAL: NCT02456012
Title: Secondary Prevention With Long-term Oral Esomeprazole for Peptic Ulcer Recurrence and Rebleeding in High-risk Rockall Scores ≥ 6 Patients
Brief Title: Long-term Oral Esomeprazole for Prevention of Peptic Ulcer Rebleeding in High-risk Patients
Acronym: Eso_1y_R6PUB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hsiu-Chi Cheng (Other)
Responsible Party: Sponsor-Investigator, Hsiu-Chi Cheng, Associate professor, National Cheng-Kung University Hospital
Organization: National Cheng-Kung University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: A-BR-104-007; R6IIT (Other: Ministry of Health and Welfare, Executive Yuan, Taiwan)
Record Dates: First submitted 2015-05-25; First posted 2015-05-28 (Estimated); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Peptic Ulcer Hemorrhage
Keywords: peptic ulcer hemorrhage; comorbidity; clinical trial
MeSH Terms: conditions — Peptic Ulcer Hemorrhage | interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- The D group (Experimental): After 3-day intravenous 8 mg/h and 16-week oral 40 mg/day esomeprazole treatment, patients receive oral esomeprazole 20 mg twice daily for 36 weeks.
  Interventions: Drug: oral esomeprazole 20 mg twice daily
- The S group (Experimental): After 3-day intravenous 8 mg/h and 16-week oral 40 mg/day esomeprazole treatment, patients receive oral esomeprazole 20 mg once daily for 36 weeks.
  Interventions: Drug: oral esomeprazole 20 mg once daily
- The C group (No Intervention): The cohort control group includes patients from a previous study who had peptic ulcer bleeding and Rockall scores ≥ 6 but who did not receive esomeprazole or other proton pump inhibitors after 3-day intravenous 8 mg/h and 16-week oral 40 mg/day esomeprazole treatment.

INTERVENTIONS:
Drug: oral esomeprazole 20 mg twice daily — for 36 weeks
  Other Names: Nexium®, 20 mg, AstraZeneca AB, Södertälje, Sweden
  Arms: The D group
Drug: oral esomeprazole 20 mg once daily — for 36 weeks
  Other Names: Nexium®, 20 mg, AstraZeneca AB, Södertälje, Sweden
  Arms: The S group

SUMMARY:
The purpose of this study is to determine whether a long-term prophylactic use of esomeprazole 20 mg twice daily or once daily has prevention effectiveness in reducing the recurrence of peptic ulcer bleeding after ulcer healed with 16-week oral esomeprazole therapy in high-risk patients whose Rockall score ≥ 6.

DETAILED DESCRIPTION:
This study is conducted at the inpatient wards of National Cheng Kung University Hospital, a tertiary health care center in Tainan, and Kaohsiung Medical University Hospital in Kaohsiung City, Taiwan. All participants give written informed consent before enrollment. Each enrolled patient receives an 80 mg loading dose of intravenous esomeprazole (Nexium®, AstraZeneca AB, Södertälje, Sweden) immediately after achieving haemostasis by gastroscopy. Patients then receive a 3-day continuous high-dose (8 mg/h) esomeprazole infusion and then receive 40 mg oral esomeprazole twice daily for 11 days and once daily for following 98 days. The total duration of intravenous and oral esomeprazole is 16 weeks. After gastroscopy to confirm enrollment eligibility and ulcer healed, all patients are assessed using the Rockall risk scoring system at the primary endoscopy. Patients with Rockall scores ≥ 6 are randomized into the double-dose (D) group or the single-dose (S) group following simple randomization procedures with a 1:1 allocation ratio according to the result by the investigator who draw an envelope from a large box of sealed envelopes each containing a written code designating the D group or the S group. Patients in the D group and S groups receive 20 mg oral esomeprazole twice daily or once daily for 36 weeks, respectively. The cohort control group includes patients from a previous study who had peptic ulcer bleeding and Rockall scores ≥ 6 but who did not receive esomeprazole or other proton pump inhibitors after 16-week proton pump inhibitor treatment.

One investigator generates the random allocation sequence and enrolls the participants and a different investigator assigns participants to interventions. The endoscopists and staff who check hemoglobin levels, hemodynamic status, melena, hematochezia or the aspirates through a nasogastric tube are blinded to the study group allocation. All enrolled patients are included in the intention-to-treat (ITT) analysis, but patients who are lost to follow-up, discontinued intervention because of adverse events, have a protocol violation or die are excluded from the per-protocol (PP) analysis of the primary endpoint.

The range of co-morbidities evaluated by the Rockall scores include disseminated malignant diseases, liver disease (liver cirrhosis, Child-Pugh A, B, or C), renal disease (end-stage renal disease, chronic kidney disease or acute kidney injury with estimated glomerular filtration rates <30 ml/min [a score of 3 for co-morbidity], or between 30 ml/min and 60 ml/min [a score of 2 for co-morbidity]), heart disease (congestive heart failure, New York Heart Association Function I to IV or coronary artery disease). Other serious co-morbidities include lung disease (chronic obstructive pulmonary disease, pulmonary tuberculosis, pneumonia or empyema), rheumatoid arthritis, sepsis, new onset cerebrovascular accident or recent history of any major surgery (on the thorax, abdomen, central nervous system, long bones or spinal bones) requiring general anesthesia within 14 days before bleeding.

The estimated rebleeding rate within 12 months in the cohort control group is about 15% based on the previous study. The investigators want to be able to detect a difference between the cohort control group and the D group, in which the rebleeding rate is proposed to be 2%, equal to patients with H. pylori ulcers after eradication. The ratio of the patient number in each experiment group (the D group and the S group) to the patient number in the control group is 2:5. With a two-side α value of 0.05 and power of 80% (β=0.20), the total number of patients required is 54 in each experiment group and 135 in the control to detect a difference between the two groups. Assuming the rate of loss follow-up is 10%, 60 patients in each experimental group are enrolled. The investigators use a nominal 0.05 rate of the p value. Data related to baseline characteristics and end points are evaluated using the Student t test, Pearson's χ2 test or Fisher's exact test and the Mann-Whitney U test. In the survival analysis, the log-rank test is used to compare the Kaplan-Meier curves among the three study groups. All tests are two-tailed and p values of less than 0.05 indicate significant differences.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants included patients ≥20 years who had undergone gastroscopy for melena, haematochezia, or haematemesis due to bleeding peptic ulcers with major stigmata of recent hemorrhage. The major stigmata of recent haemorrhage were classified as Forrest class Ia, Ib, IIa, and IIb. All of the stigmata are given one or a combination of endoscopic therapies, including local injection of diluted epinephrine 1:10000, bipolar heated probe, argon plasma coagulation, band ligation, or hemoclip therapy. Patients will undergo a follow-up endoscopy about 12 to 16 weeks later to confirm that the ulcer has healed to be less than 0.5 cm; otherwise, patients are not enrolled.

Exclusion Criteria:

* Patients are excluded if they had tumor bleeding or ulcer bleeding due to the presence of a Dieulafoy lesion or mechanical factors (e.g, gastrostomy tube induction), comorbid with reflux esophagitis grade C or D, Barrett's esophagus, or marginal ulcer bleeding, hypersensitivity to esomeprazole or any component of the formulation, or had previously participated in the study. Because of concern for patient safety with certain drug-drug interactions, patients who receive anti-platelet therapy, e.g., aspirin, clopidogrel, or others for prophylaxis of established cardiovascular or cerebrovascular diseases will be excluded.

Ages: 20 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
The recurrent peptic ulcer bleeding during the 1st year | 52 weeks
  The recurrent bleeding is deﬁned as 1) recurrent melena, haematochezia, the presence of bloody aspirates through a nasogastric tube and 2) relapse of haemodynamic instability, including systolic blood pressure <90 mm Hg, heart rate >120 bpm or a drop in haemoglobin concentration of >2 g/dL, or sudden increase in transfusion requirements. For each patient with either suspected or active rebleeding, the hemoglobin level and gastroscopy are performed to confirm any blood or coffee-ground-like materials in the stomach, or the persistence of stigmata indicating recent haemorrhage. The gastroscopy also determines whether the source of rebleeding was a peptic ulcer or some other non-ulcer bleeding source, such as varices.

SECONDARY OUTCOMES:
The recurrence of peptic ulcer confirmed by follow-up endoscopy | between the 17th and 52th weeks
  In each patient, the follow-up endoscopy will be performed during the period between the 17th and 52th weeks and the definition of recurrence of ulcer is the size of ulcer > 0.5 cm.
The recurrent peptic ulcer bleeding during the second year-and-thereafter | Since the 2nd year to the study end
  After the 52-week therapy, the patients in Group D and S used oral PPIs or not at the discretion of their physicians according to clinical needs. Thus, these patients are divided into the PPIs on-demand group and the PPIs discontinued group. The definition of recurrent bleeding is as the primary outcome.

OTHER OUTCOMES:
Medical events, including diarrhea and pneumonia, and bone fracture | During the period of taking PPIs and until two weeks after discontinuing PPIs.
  The definition of diarrhea is that the presence of loose or watery stools ≥ three times a day lasted for one day at least. The definition of pneumonia is the presence of one of the symptoms and signs of fever, chills, purulent productive cough, and shortness of breath plus a typical infiltrative patch on chest X-ray. Additionally, any bone fracture, including a partial or complete break in the bone, is monitored until the last follow-up date at outpatient departments.

CONTACTS AND LOCATIONS:
Overall Officials: Bor-Shyang Sheu, MD, Study Director — National Cheng-Kung University Hospital
Locations (1):
- Helicobacter pylori study group, National Cheng Kung University Hospital, Tainan, Taiwan

REFERENCES:
- [Background] Chan HL, Wu JC, Chan FK, Choi CL, Ching JY, Lee YT, Leung WK, Lau JY, Chung SC, Sung JJ. Is non-Helicobacter pylori, non-NSAID peptic ulcer a common cause of upper GI bleeding? A prospective study of 977 patients. Gastrointest Endosc. 2001 Apr;53(4):438-42. doi: 10.1067/mge.2001.112840. PMID 11275883
- [Background] Hung LC, Ching JY, Sung JJ, To KF, Hui AJ, Wong VW, Leong RW, Chan HL, Wu JC, Leung WK, Lee YT, Chung SC, Chan FK. Long-term outcome of Helicobacter pylori-negative idiopathic bleeding ulcers: a prospective cohort study. Gastroenterology. 2005 Jun;128(7):1845-50. doi: 10.1053/j.gastro.2005.03.026. PMID 15940620
- [Background] Chow DK, Sung JJ. Non-NSAID non-H. pylori ulcer disease. Best Pract Res Clin Gastroenterol. 2009;23(1):3-9. doi: 10.1016/j.bpg.2008.11.010. PMID 19258182
- [Background] Wong GL, Wong VW, Chan Y, Ching JY, Au K, Hui AJ, Lai LH, Chow DK, Siu DK, Lui YN, Wu JC, To KF, Hung LC, Chan HL, Sung JJ, Chan FK. High incidence of mortality and recurrent bleeding in patients with Helicobacter pylori-negative idiopathic bleeding ulcers. Gastroenterology. 2009 Aug;137(2):525-31. doi: 10.1053/j.gastro.2009.05.006. Epub 2009 May 13. PMID 19445937
- [Background] Rockall TA, Logan RF, Devlin HB, Northfield TC. Risk assessment after acute upper gastrointestinal haemorrhage. Gut. 1996 Mar;38(3):316-21. doi: 10.1136/gut.38.3.316. PMID 8675081
- [Background] Cheng HC, Wu CT, Chang WL, Cheng WC, Chen WY, Sheu BS. Double oral esomeprazole after a 3-day intravenous esomeprazole infusion reduces recurrent peptic ulcer bleeding in high-risk patients: a randomised controlled study. Gut. 2014 Dec;63(12):1864-72. doi: 10.1136/gutjnl-2013-306531. Epub 2014 Mar 21. PMID 24658598
- [Background] Marmo R, Koch M, Cipolletta L, Capurso L, Grossi E, Cestari R, Bianco MA, Pandolfo N, Dezi A, Casetti T, Lorenzini I, Germani U, Imperiali G, Stroppa I, Barberani F, Boschetto S, Gigliozzi A, Gatto G, Peri V, Buzzi A, Della Casa D, Di Cicco M, Proietti M, Aragona G, Giangregorio F, Allegretta L, Tronci S, Michetti P, Romagnoli P, Piubello W, Ferri B, Fornari F, Del Piano M, Pagliarulo M, Di Mitri R, Trallori G, Bagnoli S, Frosini G, Macchiarelli R, Sorrentini I, Pietrini L, De Stefano S, Ceglia T, Chiozzini G, Salvagnini M, Di Muzio D, Rotondano G; Italian registry on upper gastrointestinal bleeding (Progetto Nazionale Emorragie Digestive--PNED 2). Predicting mortality in non-variceal upper gastrointestinal bleeders: validation of the Italian PNED Score and Prospective Comparison with the Rockall Score. Am J Gastroenterol. 2010 Jun;105(6):1284-91. doi: 10.1038/ajg.2009.687. Epub 2010 Jan 5. PMID 20051943
- [Derived] Chiang HC, Yang EH, Hu HM, Chen WY, Chang WL, Wu CT, Wu DC, Sheu BS, Cheng HC. An extended 36-week oral esomeprazole improved long-term recurrent peptic ulcer bleeding in patients at high risk of rebleeding. BMC Gastroenterol. 2022 Oct 21;22(1):439. doi: 10.1186/s12876-022-02534-0. PMID 36271335